CLINICAL TRIAL: NCT06164977
Title: Chronic Total Coronary Occlusion Treatment Results 6 Years After Bioresorbable Scaffold Implantation
Acronym: CTO_BVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO_BVS
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Angina Pectoris; Coronary Artery Disease; Occlusion, Coronary
Keywords: Atherosclerosis; Chronic total coronary occlusion; Intravascular ultrasound; Optic coherence tomography
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease; Coronary Occlusion; Atherosclerosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Single group consists of study participants who where treated for chronic total coronary occlusion with bioresorbable scaffolds
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chronic total coronary occlusion (Other): Participants who underwent percutaneous coronary intervention for chronic total coronary occlusion revascularization with bioresorbable scaffold.
  Interventions: Procedure: Percutaneous coronary intervention.

INTERVENTIONS:
Procedure: Percutaneous coronary intervention. — Revascularization of chronic total coronary occlusion.

SUMMARY:
Aim of the study is to evaluate chronic total coronary occlusion treatment results 6 years after bioresorbable scaffold implantation by quantitative coronary analysis, intravascular ultrasound and optical coherence tomography.

DETAILED DESCRIPTION:
The study aims to assess the outcomes of treating chronic total coronary occlusion (CTO) using bioresorbable scaffolds six years after implantation. The evaluation employs quantitative coronary analysis (QCA), intravascular ultrasound (IVUS), and optical coherence tomography (OCT) as invasive imaging tools. Clinical follow-ups were conducted at one and six years post-implantation to ensure a comprehensive understanding of the long-term safety and feasibility of bioresorbable scaffold implantation for CTO.

The primary outcome measure is defined as the target lesion failure of the treated chronic total coronary occlusion segment. Target lesion failure typically encompasses a composite endpoint that includes clinical events such as cardiac death, target vessel myocardial infarction, and clinically-driven target lesion revascularization.

The use of QCA allows for the quantitative assessment of the coronary arteries, providing measurements of vessel diameter and lesion length. IVUS is employed to obtain detailed images of the vessel wall, helping to visualize the morphology of the treated segment and assess the presence of any complications such as stent malapposition or edge dissections. OCT, with its high resolution, allows for detailed imaging of the coronary artery, providing information on plaque composition and stent apposition.

By combining these invasive imaging tools with clinical follow-ups at specified intervals, the study aims to provide a comprehensive evaluation of the long-term efficacy and safety of bioresorbable scaffold implantation in the treatment of chronic total coronary occlusion. The focus on target lesion failure as the primary outcome measure ensures a clinically relevant assessment of the success of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 100% occlusion of a coronary artery for a duration of greater than or equal to 3 months based on angiographic evidence.

Exclusion Criteria:

* Participant withdrawal from study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure | 6 years
  Target Lesion Failure (TLF) will be assessed as the number of participants experiencing at least one of the following events during the follow-up period: cardiovascular death, clinically driven target lesion revascularization, target vessel myocardial infarction and stent thrombosis according to the Academic Research Consortium.

CONTACTS AND LOCATIONS:
Locations (1):
- Pauls Stradins Clinical University Hospital, Riga, Rīga, Latvia